CLINICAL TRIAL: NCT06938139
Title: Defining Benchmarks for Gastric Cancer Patients Underwent Minimal Invasive Gastrectomy: A Multicentre Analysis
Brief Title: Defining Benchmarks for Gastric Cancer Patients Underwent Minimal Invasive Gastrectomy
Status: Active, not recruiting | Type: Observational
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., Director of Gastric Surgery department, Fujian Medical University
Other Study IDs: Benchmark-MISGC
Record Dates: First submitted 2025-03-28; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Gastric Adenocarcinoma; Surgery, Laparoscopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: None-placebo — None, observational study

SUMMARY:
The Benchmark-MISGC study was a large-scale retrospective observational study launched by the China Gastric Cancer Surgical Union, aiming to establish the benchmarks of the short- and long-term outcomes for gastric cancer patients who underwent minimal invasive gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with postoperative histologically confirmed gastric adenocarcinoma at stages T1-4a, N0/+, M0;
2. underwent robotic or laparoscopic gastrectomies with curative intent

Exclusion Criteria:

1. ASA class > 3;
2. remnant gastric cancer;
3. concurrent/previous malignant disease;
4. Distant metastasis;
5. Palliative resection;
6. Abodominal exploration.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with postoperative histologically confirmed gastric adenocarcinoma at stages T1-4a, N0/+, M0 and treated with robotic or laparoscopic gastrectomies with curative intent along with lymph node dissection between January 2009 and April 2024.
Sampling Method: Non-Probability Sample
Enrollment: 90000 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Benchmark values of overall complication | 30 days
  Median values of continuous variables and the proportions of categorical variables were calculated per participating centre. Benchmark values, indicating 'best achievable' results for each outcome indicator, were set at the 25th percentile for positive parameters (for example lymph node yield) or the 75th percentile for negative parameters (for example complications) of the centers' median values. Postoperative complications were evaluated within 30 days following surgery. These postoperative complications include gastrointestinal-related complications, incision-related complications, respiratory complications, cardiovascular and cerebrovascular complications, urinary system complications, infection complications, embolism complications, and other complications. The grading of postoperative complications adopts the Clavien-Dindo classification.

SECONDARY OUTCOMES:
Benchmark values of Overall survival (OS) | 1-year, 2-year and 3-year
  Benchmark values of 1-year, 2-year and 3-year OS. OS was defined as the time from surgery to death from any cause or last follow-up.
Benchmark values of Disease-specific survival (DSS) | 1-year, 2-year, and 3-year
  Benchmark values of 1-year, 2-year and 3-year DSS. DSS was defined as the time from surgery to death from gastric cancer, or last follow-up.
benchmark value of the number of harvest lymph nodes | 1 month
  the number of harvest lymph nodes
Benchmark values of Mortality rates | 30 days
  Patient died during hospitalization.
Benchmark values of the incidence of intraoperative complications | 1 days
  Intraoperative complications were defined as bleeding due to named vessel injury, injury to visceral organs, mechanical factor-related problems, cardiopulmonary dysfunction due to hypercapnia, and other complications
Benchmark values of Intraoperative blood loss | 1 day
  Intraoperative blood loss
Benchmark values of operation time | 1 day
  From skin incision to skin closure
Benchmark values of textbook Outcome | 30 days
  Textbook outcome (TO) was defined based on review of existing TO metrics in the literature including outcomes such as complete-potentially curative status, no intraoperative complications, no eventful postoperative complications (Clavien-Dindo grade III or higher), 15 lymph nodes(LNs) examined, hospital stay < 21days, no reintervention (surgical, endoscopic or radiological) within 30 days after surgery, no readmission to the intensive care unit (ICU) within 30 days after surgery, no postoperative mortality within 30 days after surgery, and no hospital readmission within 30 days after discharge. When all nine desired health outcomes were realized, TO was achieved.

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian medical university union hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided